CLINICAL TRIAL: NCT05405777
Title: A Retrospective Study to Evaluate the Clinical Outcome According to Treatment in Atypical Hemolytic Uremic Syndrome (aHUS) Patients in South Korea
Brief Title: A Retrospective Study to Evaluate the Clinical Outcome According to Treatment in aHUS Patients in South Korea
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-ECU-501
Record Dates: First submitted 2022-05-13; First posted 2022-06-06 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: aHUS
Keywords: aHUS; eculizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective

- To determine the clinical prognosis by identifying the disease course and severity by treatment with or without eculizumab in patients with aHUS in Korea.

Secondary objectives

* To determine the clinical prognosis of the disease in all patients with aHUS in Korea.
* To determine the clinical prognosis of the disease in patients diagnosed with aHUS prior to the initiation of eculizumab reimbursement system in Korea.
* To determine the treatment responses by treatment options in patients with aHUS in Korea.
* To identify risk factors that affect mortality in all patients with aHUS in Korea.
* To investigate the recurrence and clinical prognosis in patients with aHUS in Korea when eculizumab is discontinued

DETAILED DESCRIPTION:
As a retrospective, non-interventional, multi-center study

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with the aHUS

Exclusion Criteria:

* Patients who are diagnosed with Shiga toxin-producing E. coli hemolytic-uremic syndrome (STEC-HUS).
* Patients with less than 10% in a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13 (ADAMTS-13) activity test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are clinically diagnosed with the atypical hemolytic uremic syndrome (aHUS).
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical prognosis (Renal survival) by treatment with or without eculizumab | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, or date of ESRD diagnosis, whichever came first
  Renal survival (end-stage renal disease [ESRD]-free survival)
Clinical prognosis (Overall survival) by treatment with or without eculizumab | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, whichever came first
  Overall survival (OS)

SECONDARY OUTCOMES:
Clinical prognosis (Renal survival) of all aHUS patients in Korea | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, or date of ESRD diagnosis, whichever came first
  Renal survival (ESRD-free survival)
Clinical prognosis (Overall survival) of all aHUS patients in Korea | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, whichever came first
  Overall survival (OS)
Clinical prognosis (Renal survival) of patients diagnosed with aHUS prior to the initiation of eculizumab reimbursement system in Korea | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, or date of ESRD diagnosis, whichever came first
  Renal survival (ESRD-free survival)
Clinical prognosis (Overall survival) of patients diagnosed with aHUS prior to the initiation of eculizumab reimbursement system in Korea | from the first onset date of TMA diagnosed as aHUS to the last follow up (within March 31, 2022), death, whichever came first
  Overall survival (OS)
Response rates of each treatment, compared to prior to start treatment | 3rd and 6th months
  Complete response of TMA

CONTACTS AND LOCATIONS:
Locations (1):
- Handok, Seoul, South Korea